CLINICAL TRIAL: NCT03492398
Title: A Randomized, Double-blind, Placebo-controlled Single Multiple Dosing, Dose Escalation Phase I Clinical Trial to Investigate HY209 Gel in Healthy Male Volunteers as a Possible Treatment Option for Atopic Dermatitis
Brief Title: A Phase I Study of HY209 Gel in Healthy Male Volunteers for Atopic Dermatitis
Acronym: Shaperon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaperon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HY209-202
Record Dates: First submitted 2018-02-15; First posted 2018-04-10 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-03

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: A randomized, double blind, placebo-controlled, single and multiple dosing, dose escalation study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort A HY209 0.05% gel (Experimental): single dose of HY209 0.05% gel or single dose of placebo
  Interventions: Drug: HY209
- Cohort A HY209 0.1% gel (Experimental): single dose of HY209 0.1% gel or single dose of placebo
  Interventions: Drug: HY209
- Cohort A HY209 0.3% gel (Experimental): single dose of HY209 0.3% gel or single dose of placebo
  Interventions: Drug: HY209
- Cohort A HY209 0.5% gel (Experimental): single dose of HY209 0.5% gel or single dose of placebo
  Interventions: Drug: HY209
- Cohort B HY209 0.1% gel (Experimental): multiple dose of HY209 0.1% gel or multiple dose of placebo
  Interventions: Drug: HY209
- Cohort B HY209 0.3% gel (Experimental): multiple dose of HY209 0.3% gel or multiple dose of placebo
  Interventions: Drug: HY209
- Cohort B HY209 0.5% gel (Experimental): multiple dose of HY209 0.5% gel or multiple dose of placebo
  Interventions: Drug: HY209

INTERVENTIONS:
Drug: HY209 — 6 subjects will be assigned to drug (HY209) and 2 subjects will be assigned to placebo.
  Other Names: HY209 gel

SUMMARY:
A randomized, double-blind, placebo-controlled single and multiple dosing, dose escalation phase I clinical trial to investigate the safety/tolerability and pharmacokinetics of HY209 gel after transdermal administration in healthy male volunteers as a possible treatment option for atopic dermatitis

DETAILED DESCRIPTION:
A composition containing G Protein Coupled Receptor 19(GPCR19) agonist HY209 and a derivative thereof is found to have a considerable effect in the treatment of atopic dermatitis and is proposed as a pharmaceutical ingredient for prevention, treatment and improvement of atopic dermatitis. The GPCR19 agonist, HY209, is superior to conventional steroid ointment and immunosuppressant ointment in the treatment and improvement of allergic dermatitis. It directly reduces the amount of serum immunoglobulin E, which is a major factor of allergic dermatitis, It increases the T helper type 1(TH1) cytokines that alleviate allergic dermatitis pathologies, reduces the T helper type 2(TH2) cytokines that aggravate allergic dermatitis pathologies, and reduces the infiltration of mast cells, eosinophils and neutrophils into the dermal cells. Thus it can be utilized as a therapeutic drug composition for atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged from 20 to 50 at screening test
* Weight 45kg ~ 90kg with BMI 17kg/m2 ~ 27kg/m2
* No skin diseases, no skin damages(scars, tattoo, etc), no hairy skin

Exclusion Criteria:

* Those who have a history of hypersensitivity or clinically significant hypersensitivity reactions to generic drugs (aspirin, antibiotics, etc.)
* Those who have clinically significant liver, kidney, respiratory, endocrine, neurologic diseases or hematologic diseases, mental diseases, especially hemorrhagic diseases (hemophilia, von Willebrand disease, etc.), cardiovascular diseases (coronary artery disease, Congestive heart failure, arrhythmia, cerebrovascular disease, etc.) or who have a history of those diseases
* Those who had clinical symptoms suspected of acute infectious disease within 2 weeks before the scheduled date of the first administration, or whose temperature measured by the screening test (eardrum) was 38.0 ° C or higher
* Those who have taken any prescription drugs, herbal medicines, crude drugs within 2 weeks before the scheduled date of administration of the medicines for clinical trials , or over-the-counter medicines or vitamin preparations within 1 week.
* Those who have a history of substance abuse, or positive urine screening tests (cannabinoid, opiates, amphetamine, cocaine, barbiturate, benzodiazepine)
* Those who have a history of smoking within 3 months (However, if they quit smoking three months before the first scheduled medication, they are eligible for selection)
* Those who have been found to be positive in serological tests (HBs antigen, hepatitis C virus antibody and HIV antibody)
* Those who drink continuously (above 21 units / week, 1 unit = 10 g of pure alcohol)
* Those who have been taking medicines by participating in other clinical trials or bioequivalence studies within 3 months prior to the date of first dosing
* Those who have been bleeding, blood drawings or blood donation of 400mL or more within 8 weeks before the scheduled date of administration of the drug for clinical trials
* Those who have vital signs measured at sitting position after the break for more than 3 minutes,

  * Low blood pressure (systolic blood pressure <90 mmHg, diastolic blood pressure <50 mmHg)
  * High blood pressure (systolic blood pressure greater than 150 mmHg, diastolic blood pressure greater than 100 mmHg)
* Test subjects who are deemed unsuitable for participating in clinical trials due to clinical laboratory tests, ECG results, or other reasons

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyungsang Yu, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A HY209 Placebo: single dose of placebo
  total 8 subjects participated.
- Cohort A HY209 0.05% Gel: single dose of HY209 0.05% gel
  total 6 subjects participated.
- Cohort A HY209 0.1% Gel: single dose of HY209 0.1% gel
  total 6 subjects participated.
- Cohort A HY209 0.3% Gel: single dose of HY209 0.3% gel
  total 6 subjects participated.
- Cohort A HY209 0.5% Gel: single dose of HY209 0.5% gel
  total 6 subjects participated.
- Cohort B Placebo: multiple dose of placebo
  total 6 subjects participated.
- Cohort B HY209 0.1% Gel: multiple dose of HY209 0.1% gel
  total 6 subjects participated.
- Cohort B HY209 0.3% Gel: multiple dose of HY209 0.3% gel
  total 6 subjects participated.
- Cohort B HY209 0.5% Gel: multiple dose of HY209 0.5% gel
  total 6 subjects participated.
Period: Overall Study
Arm/Group | Cohort A HY209 Placebo | Cohort A HY209 0.05% Gel | Cohort A HY209 0.1% Gel | Cohort A HY209 0.3% Gel | Cohort A HY209 0.5% Gel | Cohort B Placebo | Cohort B HY209 0.1% Gel | Cohort B HY209 0.3% Gel | Cohort B HY209 0.5% Gel
Started | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A Placebo: single dose of placebo 8 subjects
- Cohort A HY209 0.05% Gel: single dose of HY209 0.05% gel 6 subjects
- Cohort A HY209 0.1% Gel: single dose of HY209 0.1% gel 6 subjects
- Cohort A HY209 0.3% Gel: single dose of HY209 0.3% gel 6 subjects
- Cohort A HY209 0.5% Gel: single dose of HY209 0.5% gel 6 subjects
- Cohort B Placebo: multiple dose of placebo 6 subjects
- Cohort B HY209 0.1% Gel: multiple dose of HY209 0.1% gel 6 subjects
- Cohort B HY209 0.3% Gel: multiple dose of HY209 0.3% gel 6 subjects
- Cohort B HY209 0.5% Gel: multiple dose of HY209 0.5% gel 6 subjects
- Total: Total of all reporting groups
Arm/Group | Cohort A Placebo | Cohort A HY209 0.05% Gel | Cohort A HY209 0.1% Gel | Cohort A HY209 0.3% Gel | Cohort A HY209 0.5% Gel | Cohort B Placebo | Cohort B HY209 0.1% Gel | Cohort B HY209 0.3% Gel | Cohort B HY209 0.5% Gel | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 56
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events
Description: Number of participants with abnormal laboratory values and/or adverse events that are related to treatment
Time Frame: upto Day 8(single dosing), upto Day 38(multiple dosing)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A Placebo: single dose of placebo
  total 8 subjects assigned.
- Cohort A HY209 0.05% Gel: single dose of HY209 0.05% gel
  total 6 subjects assigned.
- Cohort A HY209 0.1% Gel: single dose of HY209 0.1% gel
  total 6 subjects assigned.
- Cohort A HY209 0.3% Gel: single dose of HY209 0.3% gel
  total 6 subjects assigned.
- Cohort A HY209 0.5% Gel: single dose of HY209 0.5% gel
  total 6 subjects assinged.
- Cohort B Placebo: multiple dose of placebo
  total 6 subjects assigned.
- Cohort B HY209 0.1% Gel: multiple dose of HY209 0.1% gel
  total 6 subjects assigned.
- Cohort B HY209 0.3% Gel: multiple dose of HY209 0.3% gel
  total 6 subjects assigned.
- Cohort B HY209 0.5% Gel: multiple dose of HY209 0.5% gel
  total 6 subjects assigned.
Arm/Group | Cohort A Placebo | Cohort A HY209 0.05% Gel | Cohort A HY209 0.1% Gel | Cohort A HY209 0.3% Gel | Cohort A HY209 0.5% Gel | Cohort B Placebo | Cohort B HY209 0.1% Gel | Cohort B HY209 0.3% Gel | Cohort B HY209 0.5% Gel
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 4 | 2 | 2 | 1 | 0 | 2 | 2 | 2 | 3

ADVERSE EVENTS:
Time Frame: upto Day 8(single dosing), upto Day 38(multiple dosing)
Description: Number of participants with abnormal laboratory values and/or adverse events that are related to treatment
Groups:
- Cohort A HY209 Placebo: single dose of placebo
  total 8 subjects assigned.
- Cohort A HY209 0.5% Gel: single dose of HY209 0.5% gel
  total 6 subjects assigned.
- Cohort B HY209 0.3% Gel: multiple dose of HY209 0.3%
  total 6 subjects assigned.
- Cohort B HY209 0.5% Gel: multiple dose of HY209 0.5%
  total 6 subjects assigned.
Arm/Group | Cohort A HY209 Placebo | Cohort A HY209 0.05% Gel | Cohort A HY209 0.1% Gel | Cohort A HY209 0.3% Gel | Cohort A HY209 0.5% Gel | Cohort B Placebo | Cohort B HY209 0.1% Gel | Cohort B HY209 0.3% Gel | Cohort B HY209 0.5% Gel
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 2/6 | 1/6 | 1/6 | 0/6 | 1/6 | 0/6 | 1/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A HY209 Placebo (N=8) | Cohort A HY209 0.05% Gel (N=6) | Cohort A HY209 0.1% Gel (N=6) | Cohort A HY209 0.3% Gel (N=6) | Cohort A HY209 0.5% Gel (N=6) | Cohort B Placebo (N=6) | Cohort B HY209 0.1% Gel (N=6) | Cohort B HY209 0.3% Gel (N=6) | Cohort B HY209 0.5% Gel (N=6)
Application site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Appication site irritation (General disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Application site pruritus (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-01-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT03492398/Prot_000.pdf